CLINICAL TRIAL: NCT00003852
Title: Phase II Study of Intensive Chemotherapy With Autologous Peripheral Blood Stem Cell Support in Patients With Cisplatin Resistant Germ Cell Tumors
Brief Title: Combination Chemotherapy Plus Peripheral Stem Cell Transplantation in Treating Patients With Germ Cell Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of patient inclusion
Sponsor: UNICANCER (Other)
Purpose: Treatment
Other Study IDs: CDR0000067015; FRE-FNCLCC-GETUG-04; EU-99004
Record Dates: First submitted 1999-11-01; First posted 2004-01-27 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Childhood Germ Cell Tumor; Extragonadal Germ Cell Tumor; Ovarian Cancer; Testicular Germ Cell Tumor
Keywords: recurrent malignant testicular germ cell tumor; childhood germ cell tumor; recurrent ovarian germ cell tumor; extragonadal germ cell tumor
MeSH Terms: conditions — Ovarian Neoplasms; Testicular Germ Cell Tumor; Testicular Neoplasms | interventions — Filgrastim; Carboplatin; Cyclophosphamide; Epirubicin; Etoposide; Ifosfamide; Paclitaxel; Thiotepa; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: cyclophosphamide
Drug: epirubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Drug: paclitaxel
Drug: thiotepa
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow patients to tolerate higher doses of chemotherapy and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy and peripheral stem cell transplantation in treating patients who have germ cell tumors that have not responded to previous chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the complete response rate (chemotherapy complete response, pathological complete response, or surgical complete response) to intensive chemotherapy with autologous peripheral blood stem cell support in patients with cisplatin resistant germ cell tumors. II. Determine duration of complete response and survival of these patients after this therapy. III. Determine the toxic effects of this regimen in these patients. IV. Determine the pharmacokinetics of this regimen and the relationship between these pharmacokinetics, nature and duration of response to treatment, and the toxic effects in these patients.

OUTLINE: This is an open label, multicenter study. Patients receive epirubicin IV over 15 minutes and paclitaxel IV over 3 hours on day 1, then filgrastim (G-CSF) subcutaneously (SQ) on days 5-14. Peripheral blood stem cells (PBSC) are collected on days 13 and 14. This course is repeated beginning on day 15. Patients then undergo a three part intensification regimen. Part I: Patients receive cyclophosphamide IV and thiotepa IV by continuous infusion on days 34 and 35. PBSC are reinfused on day 38, and G-CSF SQ is administered from day 39 until blood cell counts recover. Part II: Patients receive etoposide IV over 2 hours, ifosfamide IV over 4 hours, and carboplatin IV over 6 hours on days 62-66. PBSC are reinfused on day 70, and eventually G-CSF begins on day 71. Part III: Patients receive etoposide, ifosfamide, and carboplatin on days 90-94 as in part II. PBSC are reinfused on day 98 and eventually G-CSF begins on day 99. Patients are followed every month for the first year, every 2 months for the second year, every 6 months for the third and fourth years, then annually thereafter.

PROJECTED ACCRUAL: A total of 45 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven germ cell tumor Seminoma or nondysgerminoma origin Gonadal (testicular or ovarian) OR Extragonadal OR Retroperitoneal OR Primitive mediastinal AFP elevated and/or HCG greater than 200 mIU/mL No growing teratoma Refractory disease to any treatment line Refractory disease is defined by the elevation of AFP and/or HCG during the chemotherapy Refractory to treatment line consisting of one conventional dose of cisplatin (dose intensity greater than 33 mg/m2/week) OR at least 1 month since last course of chemotherapy with or without increase in the size of measurable lesions OR Received 2 regimens of conventional chemotherapy, typically the following: Bleomycin, etoposide, and cisplatin: 3-4 courses* OR Etoposide and cisplatin: 4 courses* AND Vinblastine, etoposide, ifosfamide, cisplatin: 4 courses of 3 week regimen (as standard salvage chemotherapy)* * Unless patients could be treated with a first line conventional treatment OR a first salvage conventional treatment especially patients who could be treated with T93 good prognosis protocol or T93 bad prognosis protocol or IT94 protocol Bidimensionally measurable disease OR Significant elevation of tumor markers: HCG, free beta-HCG, AFP OR Evaluable disease plus increase in tumor markers No germ cell CNS tumors or clinically significant CNS metastases

PATIENT CHARACTERISTICS: Age: Over 15 Performance status: ECOG 0-2 Life expectancy: Greater than 3 months Hematopoietic: WBC greater than 3,000/mm3 AND Platelet count greater than 150,000/mm3 Hepatic: Bilirubin less than 1.5 times normal SGOT/SGPT less than 2 times upper limit of normal (ULN) Alkaline phosphatase less than 2 times ULN Gamma glutamyl transferase less than 2 times ULN Renal: Creatinine less than 1.4 mg/dL Creatine clearance greater than 60 mL/min Cardiovascular: No cardiac insufficiency LVEF at least 50% Other: HIV negative No other malignancy except basal cell skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No prior intensive chemotherapy with stem cell support Endocrine therapy: Not specified Radiotherapy: Prior prophylactic anterior irradiation of the diaphragm for stage I seminoma allowed Surgery: Not specified

Ages: 15 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 1998-03; Primary Completion 2000-03 (Actual); Study Completion 2000-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Biron, MD, Study Chair — Centre Leon Berard
Locations (18):
- France (18):
  - Centre Paul Papin, Angers
  - CHR de Besancon - Hopital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Centre Regional Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Lute Contre le Cancer,Georges-Francois Leclerc, Dijon
  - CHR de Grenoble - La Tronche, Grenoble
  - Clinique Saint Michel, La Rochelle
  - Centre Leon Berard, Lyon
  - Institut J. Paoli and I. Calmettes, Marseille
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hopital d'Instruction des Armees du Val de Grace, Paris
  - Institut Jean Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - Centre Rene Huguenin, Saint-Cloud
  - Hopitaux Universitaire de Strasbourg, Strasbourg
  - Institut Gustave Roussy, Villejuif